CLINICAL TRIAL: NCT01736254
Title: Effect of Gemfibrozil on the Pharmacokinetics of Evacetrapib (LY2484595) in Healthy Subjects
Brief Title: A Study of Evacetrapib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14701; I1V-MC-EIBD (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — evacetrapib; Gemfibrozil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gemfibrozil (Experimental): Single oral dose of 600 milligrams (mg) gemfibrozil on Day 1
  Interventions: Drug: Gemfibrozil
- Evacetrapib (Experimental): Oral doses of 130 mg evacetrapib once a day (QD) for 10 days (Day 2 through Day 12)
  Interventions: Drug: Evacetrapib
- Evacetrapib + Gemfibrozil (Experimental): Oral doses of 600 mg gemfibrozil twice a day (BID) and 130 mg evacetrapib QD for 10 days (Day 13 through Day 22). Single oral dose of 600 mg gemfibrozil on Day 23.
  Interventions: Drug: Evacetrapib; Drug: Gemfibrozil

INTERVENTIONS:
Drug: Evacetrapib
  Other Names: LY2484595
  Arms: Evacetrapib; Evacetrapib + Gemfibrozil
Drug: Gemfibrozil
  Arms: Evacetrapib + Gemfibrozil; Gemfibrozil

SUMMARY:
The purpose of this study is to determine whether concentrations of the study drug (evacetrapib) in the blood stream is the same or is different when the person is also taking gemfibrozil (a drug used to lower lipid levels). Each participant will receive gemfibrozil alone, evacetrapib alone, and both drugs in combination. There is no washout period between doses. The safety of both of the study drugs given together will be evaluated. Information about any side effects that may have occurred will also be collected. This study will last approximately 36 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants as determined by medical history and physical examination
* Have a body mass index of 18 to 32 kilograms per square meter (kg/m^2)

Exclusion Criteria:

* Have known allergies to evacetrapib and gemfibrozil, related compounds or any components of the formulation
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Currently smoke cigarettes or use tobacco or nicotine substitutes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All participants were assigned to the following treatment regimen:
  Period 1: Single oral dose of 600 milligrams (mg) gemfibrozil in the morning of Day 1.
  Period 2: Oral doses of 130 mg evacetrapib once a day (QD) for 11 days (Days 2 to 12).
  Period 3: Oral doses of 600 mg gemfibrozil twice a day (BID) and 130 mg evacetrapib QD for 10 days (Days 13 to 22), with a single dose of 600 mg gemfibrozil on Day 23.
Period: Period 1 (Day 1)
Arm/Group | All Participants
Started | 24
Received at Least One Dose of Study Drug | 24
Completed | 24
Not Completed | 0
Period: Period 2 (Days 2 to 12)
Arm/Group | All Participants
Started | 24
Completed | 21
Not Completed | 3
Not completed — Adverse Event | 3
Period: Period 3 (Days 13 to 23)
Arm/Group | All Participants
Started | 21
Completed | 20
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- All Participants: All participants were assigned to the following treatment regimen:
  Period 1: Single oral dose of 600 mg gemfibrozil in the morning of Day 1.
  Period 2: Oral doses of 130 mg evacetrapib QD for 11 days (Days 2 to 12).
  Period 3: Oral doses of 600 mg gemfibrozil BID and 130 mg evacetrapib QD for 10 days (Days 13 to 22), with a single dose of 600 mg gemfibrozil on Day 23.
Arm/Group | All Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14
  Black | 7
  Multiple | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Evacetrapib
Description: Venous blood samples were taken on Day 11 for PK parameter estimates of evacetrapib alone and on Day 22 for PK parameter estimates of evacetrapib when coadministered with gemfibrozil.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours postdose on Day 11 and Day 22
Population: All participants who received at least 1 dose of evacetrapib or gemfibrozil and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- Evacetrapib: Oral doses of 130 mg evacetrapib QD for 10 days (Day 2 through Day 12).
- Evacetrapib + Gemfibrozil: Oral doses of 600 mg gemfibrozil BID and 130 mg evacetrapib QD for 10 days (Day 13 through Day 22). Single oral dose of 600 mg gemfibrozil on Day 23.
Arm/Group | Evacetrapib | Evacetrapib + Gemfibrozil
Number analyzed (Participants) | 22 | 20
nanograms/milliliter (ng/mL) | 1270 (26) | 1290 (26)

2. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve Over a 24 Hour Dosing Interval (AUCτ) of Evacetrapib
Description: as for outcome 1
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours postdose on Day 11 and Day 22
Population: All participants who received at least 1 dose of evacetrapib or gemfibrozil and had evaluable AUCτ data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliliter (ng*h/mL)
Arm/Group | Evacetrapib | Evacetrapib + Gemfibrozil
Number analyzed (Participants) | 22 | 19
nanograms*hours/milliliter (ng*h/mL) | 11300 (20) | 11400 (21)

3. Primary Outcome: Pharmacokinetics (PK): Time of Maximum Observed Drug Concentration (Tmax) of Evacetrapib
Description: as for outcome 1
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours postdose on Day 11 and Day 22
Population: All participants who received at least 1 dose of evacetrapib or gemfibrozil and had evaluable Tmax data.
Measure: Median (Full Range); unit: hours
Arm/Group | Evacetrapib | Evacetrapib + Gemfibrozil
Number analyzed (Participants) | 22 | 20
hours | 4.00 [2.02 to 6.00] | 3.00 [2.00 to 4.00]

4. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve Over a 12 Hour Dosing Interval (AUCτ) of Gemfibrozil
Description: Venous blood samples were taken on Day 1 for PK parameter estimates of gemfibrozil alone and on Day 13 for PK parameter estimates of gemfibrozil when coadministered with evacetrapib.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose on Day 1 and Day 13
Population: All participants who received at least 1 dose of evacetrapib or gemfibrozil and had evaluable AUCτ data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Gemfibrozil: Single oral dose of 600 mg gemfibrozil on Day 1.
Arm/Group | Gemfibrozil | Evacetrapib + Gemfibrozil
Number analyzed (Participants) | 24 | 21
ng*h/mL | 55700 (23) | 53800 (22)

5. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Gemfibrozil
Description: as for outcome 4
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose on Day 1 and Day 13
Population: All participants who received at least 1 dose of evacetrapib or gemfibrozil and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Gemfibrozil | Evacetrapib + Gemfibrozil
Number analyzed (Participants) | 24 | 21
ng/mL | 17400 (32) | 16800 (34)

6. Secondary Outcome: Pharmacokinetics (PK): Time of Maximum Observed Drug Concentration (Tmax) of Gemfibrozil
Description: as for outcome 4
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose on Day 1 and Day 13
Population: All participants who received at least 1 dose of evacetrapib or gemfibrozil and had evaluable Tmax data.
Measure: Median (Full Range); unit: hours
Arm/Group | Gemfibrozil | Evacetrapib + Gemfibrozil
Number analyzed (Participants) | 24 | 21
hours | 1.00 [1.00 to 4.00] | 1.08 [1.08 to 4.00]

ADVERSE EVENTS:
Arm/Group | Gemfibrozil | Evacetrapib | Evacetrapib + Gemfibrozil
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 1/24 | 8/24 | 7/21
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemfibrozil (N=24) | Evacetrapib (N=24) | Evacetrapib + Gemfibrozil (N=21)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Bowel movement irregularity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days